CLINICAL TRIAL: NCT04644809
Title: A Single-Ascending and Repeat-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3561774
Brief Title: A Study of LY3561774 in Participants With Dyslipidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17825; J3F-MC-EZCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-24; First posted 2020-11-25 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08-01

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3561774 (Part A) (Experimental): Single ascending doses of LY3561774 administered subcutaneously (SC).
  Interventions: Drug: LY3561774
- LY3561774 (Part B) (Experimental): Repeat doses of LY3561774 administered SC.
  Interventions: Drug: LY3561774
- LY3561774 (Part C) (Experimental): Single doses of LY3561774 administered SC in Japanese Participants.
  Interventions: Drug: LY3561774
- Placebo (Part A, B & C) (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3561774 — Administered SC.
  Arms: LY3561774 (Part A); LY3561774 (Part B); LY3561774 (Part C)
Drug: Placebo — Administered SC.
  Arms: Placebo (Part A, B & C)

SUMMARY:
This is a 3-part study. In Parts A and B, the main purpose is to evaluate the safety and tolerability of the study drug known as LY3561774 in participants with dyslipidemia (high blood fat levels). How the body processes the study drug and the effect of the study drug on blood fat levels will also be investigated. Part C will mainly evaluate the safety and tolerability of LY3561774 as well as how the body processes the study drug in Japanese participants. The study may last up 52, 56 and 28 weeks for each participant in Parts A, B and C, respectively. There are up to 22, 26 and 16 visits in Parts A, B and C, respectively.

ELIGIBILITY:
Inclusion Criteria:

* For Parts A and B, have a fasting triglyceride (TG) level greater than or equal to (≥) 150 milligram/deciliter (mg/dL) and less than 500 mg/dL, as well as low density lipoprotein cholesterol (LDL-C) level greater than or equal to (≥) 70 mg/dL
* For Part C, participants should be first-generation Japanese origin.
* Have a body mass index (BMI) of 18.5 to 40.0 kilograms per square meter (kg/m²)
* Male participants must agree to adhere to contraception restrictions and female participants must not be able to get pregnant

Exclusion Criteria:

* Have taken any prescription medications that are for lowering serum TGs within the past 2 months (use of statins is allowed if the dose has been stable for 8 weeks)
* Have Type 1 diabetes
* Are currently participating in or completed a clinical trial within the last 30 days
* Are heavy alcohol drinkers or heavy cigarette smokers
* Have donated blood of more than 500 millilitres (mL) in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 53
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve from Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of LY3561774 | Predose through Day 8
  PK: AUC[0-tlast] of LY3561774
PK: Maximum Observed Drug Concentration (Cmax) of LY3561774 | Predose through Day 8
  PK: Cmax of LY3561774
PK: Time of Maximum Observed Concentration (Tmax) of LY3561774 | Predose through Day 8
  PK: Tmax of LY3561774
PD: Change From Baseline in Fasting Triglyceride (TG) and low-density lipoprotein cholesterol (LDL-C) | Predose through Week 53
  PD: Change From Baseline in Fasting TG and LDL-C

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Qps-Mra, Llc, South Miami, Florida
  - Hassman Research Institute, Marlton, New Jersey
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ray KK, Linnebjerg H, Michael LF, Shen X, Ma X, Lim S, Zhen EY, Dudek H, Abrams M, Saxena U, Turanov A, Nicholls SJ, Ruotolo G. Effect of ANGPTL3 Inhibition With Solbinsiran in Preclinical and Early Human Studies. J Am Coll Cardiol. 2025 May 20;85(19):1803-1818. doi: 10.1016/j.jacc.2025.03.005. Epub 2025 Mar 30. PMID 40158211
- See also: A Study of LY3561774 in Participants With Dyslipidemia — https://trials.lillytrialguide.com/en-US/trial/6o9PZPIhCp7DEVhxSrEnhY